CLINICAL TRIAL: NCT03013062
Title: Derivation of New Formula Relating Pulmonary Acceleration Time and Mean Pulmonary Artery Pressure in Indian Population and Comparison With Previous Formulas
Brief Title: Relation Between Mean Pulmonary Artery Pressure and Pulmonary Acceleration Time and Comparison With Previous Formulae
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Ganesh Kumar Munirathinam, Fellow resident, Department of anesthesia and intensive care, Principal investigator, Post Graduate Institute of Medical Education and Research, Chandigarh
Other Study IDs: INT/IEC/2016/2641
Record Dates: First submitted 2017-01-02; First posted 2017-01-06 (Estimated); Last update posted 2017-06-02 (Actual); Status verified 2017-06

CONDITIONS: Pulmonary Hypertension
MeSH Terms: conditions — Hypertension, Pulmonary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- WITH PULMONARY HYPERTENSION: It is defined as MPAP > 25 mm Hg at rest or >30 mm Hg during exercise with PVR > 3 wood units and PCWP < 15 mm Hg.

SUMMARY:
Since the pulmonary artery hypertension is defined based on MPAP and the two previous formulae relating MPAP and PAT were derived in western population, the investigator planned to conduct a prospective study to derive a new formula for measuring MPAP from PAT in Indian population and compare the accuracy of all the three formulae

DETAILED DESCRIPTION:
After obtaining ethics committee approval and informed patient consent, minimum 25 patients > 18 years of age who are undergoing cardiac surgery with the invasive monitoring of pulmonary artery pressure will be enrolled in this study.The demographics and the preoperative echocardiographic measurement will be noted. In the operating room, once the intravenous access is obtained, central venous catheterisation and pulmonary artery catheterisation will be done as per the institutional protocol. Once the Transthoracic echocardiogram (TTE) is performed patient will be induced with opioids, intravenous or inhalational agents, and muscle relaxant according to the patient clinical and hemodynamic condition. Once the patient airway is secured with tracheal tube, transesophageal echocardiogram (TEE) will be performed before and after bypass, which is routine in all patients undergoing cardiac surgery in the institution. Echocardiographic images will be analysed by two separate echocardiographers to detect inter-individual variability. Patient blood pressure and heart rate will be maintained within 20% of their baseline value throughout surgery. Based on the patient condition at the end of surgery, extubation will be done in the operating room or in intensive care unit (ICU) after a period of elective ventilation.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age who are undergoing cardiac surgery with the invasive monitoring of pulmonary artery pressure

Exclusion Criteria:

* Patients with known right ventricular outflow tract obstruction, intra-cardiac shunt lesions will be excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: > 18 years of age who are undergoing cardiac surgery with the invasive monitoring of pulmonary artery pressure
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2017-01; Primary Completion 2017-06 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Pulmonary acceleration time | Till post-extubation, an average of 2 days

CONTACTS AND LOCATIONS:
Overall Officials: GANESH KUMAR M, Principal Investigator — PGIMER, CHANDIGARH
Locations (1):
- PGIMER, Chandigarh, India